CLINICAL TRIAL: NCT00682422
Title: Kid STRIDE: Exploring Participation in a Family-based Intervention
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Other Study IDs: M-2007-1471
Record Dates: First submitted 2008-05-16; First posted 2008-05-22 (Estimated); Last update posted 2015-10-05 (Estimated); Status verified 2010-06

CONDITIONS: Obesity
Keywords: pediatrics, overweight, obese, behavioral intervention
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Parent & Child Dyad

SUMMARY:
The aim of this qualitative study is to explore parental and child perceptions of participating in a family-based behavioral intervention targeting healthy behaviors.

DETAILED DESCRIPTION:
Children ages 9-14 have been participating in the Kid STRIDE study which is a family-based behavioral intervention for obese children. Participants will be divided into 3 groups according to their change in weight: 1) children who lost greater than 5% of body weight; 2) children who lost less than 5% of body weight or gained less than 1% of body weight; 3) children who gained greater than 1% of body weight. We will invite five families from each of groups 1 and 3 to participate in an open-ended interview.

ELIGIBILITY:
Inclusion Criteria:

* Completed the 15-week primary intervention phase of Kid STRIDE

Ages: 9 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Participants in the current Kid STRIDE behavioral intervention study.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2008-02; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Explore parental and child perceptions of participating in a family-based behavioral intervention targeting weight reduction. | After completion of primary group intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Ellen R Wald, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

REFERENCES:
- [Background] Whitlock EP, Williams SB, Gold R, Smith PR, Shipman SA. Screening and interventions for childhood overweight: a summary of evidence for the US Preventive Services Task Force. Pediatrics. 2005 Jul;116(1):e125-44. doi: 10.1542/peds.2005-0242. PMID 15995013
- [Background] Ogden CL, Flegal KM, Carroll MD, Johnson CL. Prevalence and trends in overweight among US children and adolescents, 1999-2000. JAMA. 2002 Oct 9;288(14):1728-32. doi: 10.1001/jama.288.14.1728. PMID 12365956
- [Background] Guo SS, Roche AF, Chumlea WC, Gardner JD, Siervogel RM. The predictive value of childhood body mass index values for overweight at age 35 y. Am J Clin Nutr. 1994 Apr;59(4):810-9. doi: 10.1093/ajcn/59.4.810. PMID 8147324
- [Background] Freedman DS, Khan LK, Serdula MK, Dietz WH, Srinivasan SR, Berenson GS. The relation of childhood BMI to adult adiposity: the Bogalusa Heart Study. Pediatrics. 2005 Jan;115(1):22-7. doi: 10.1542/peds.2004-0220. PMID 15629977
- [Background] Strauss RS. Childhood obesity and self-esteem. Pediatrics. 2000 Jan;105(1):e15. doi: 10.1542/peds.105.1.e15. PMID 10617752
- [Background] Golan M. Parents as agents of change in childhood obesity--from research to practice. Int J Pediatr Obes. 2006;1(2):66-76. doi: 10.1080/17477160600644272. PMID 17907317